CLINICAL TRIAL: NCT05760599
Title: Candonilimab Plus Bevacizumab as Second-line Treatment for Patients With Advanced Hepatocellular Carcinoma Who Progressed on Atezolizumab Plus Bevacizumab: a Single Arm, Phase 2 Trial
Brief Title: Candonilimab Plus Bevacizumab for Patients With Advanced HCC Who Progressed on A+T
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shi Ming (Other)
Responsible Party: Sponsor-Investigator, Shi Ming, Proffessor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S104B
Record Dates: First submitted 2023-02-26; First posted 2023-03-08 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-02

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Candonilimab Plus Bevacizumab; Atezolizumab Plus Bevacizumab
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Candonilimab Plus Bevacizumab (Experimental): Candonilimab 10mg/kg, Bevacizumab 15mg/kg, every 3 week
  Interventions: Drug: Candonilimab; Drug: Bevacizumab

INTERVENTIONS:
Drug: Candonilimab — 10mg/kg, iv.drip, every 3 week
Drug: Bevacizumab — 15mg/kg, iv.drip, every 3 week

SUMMARY:
To explore the efficacy and safety of candonilimab plus bevacizumab for patients with advanced hepatocellular carcinoma who progressed on atezolizumab plus bevacizumab.

DETAILED DESCRIPTION:
Atezolizumab plus bevacizumab is the first-line treatent for patients with advanced hepatocellular carcinoma. However, the second-line treatment is absent for patients who progressed on atezolizumab plus bevacizumab. Candonilimab is a humanized bisspecific monoclonal antibody against PD-1/ CTLA-4 IgG1. Candonilimab plus lenvatinib showed strong anti-tumor effect, with objective response of 44%. This single-arm, prospective, phase 2 trial is to explore the efficacy and safety of candonilimab plus bevacizumab for patients with advanced hepatocellular carcinoma who progressed on atezolizumab plus bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of HCC was based on the diagnostic criteria for HCC used by the European Association for the Study of the Liver (EASL)
* Patients must have at least one tumor lesion that can be accurately measured according to EASL criteria.
* Barcelona clinic liver cancer-stage C
* Eastern Cooperative Oncology Group performance status of 0 to 2
* Patients have received atezolizumab plus bevacizumab and the tumor have progressed. Patients have not received other treatmets except for the atezolizumab plus bevacizumab.
* No Cirrhosis or cirrhotic status of Child-Pugh class A only
* Not amendable to surgical resection ,local ablative therapy and any other cured treatment.
* The following laboratory parameters:

Hemoglobin ≥ 8.5 g/dL Total bilirubin ≤ 30mmol/L Serum albumin ≥ 32 g/L ASL and AST ≤ 5 x upper limit of normal Serum creatinine ≤ 1.5 x upper limit of normal INR ≤ 1.5 or PT/APTT within normal limits Absolute neutrophil count (ANC) >1,500/mm3

• Ability to understand the protocol and to agree to and sign a written informed consent document

Exclusion Criteria:

* Evidence of hepatic decompensation including ascites, gastrointestinal bleeding or hepatic encephalopathy
* Known history of HIV
* History of organ allograft
* Known or suspected allergy to the investigational agents or any agent given in association with this trial.
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* Evidence of bleeding diathesis.
* Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry.
* Known central nervous system tumors including metastatic brain disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-02-27 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
DCR per RECIST 1.1 | 12 months
  DCR （Disease Control Rate） include complete response, partial response and stable Disease per RECIST 1.1

SECONDARY OUTCOMES:
Overall survival (OS) | 12 months
  OS is the length of time from the date of randomization until death from any cause.
Progression free survival (PFS) | 12 months
  PFS is defined as the time from the date of randomization to the date of the first objectively documented tumor progression or death due to any cause.
ORR per RECIST 1.1 | 12 months
  Objective response rate (complete response+partial response) per RECIST 1.1
Adverse events | 30 days
  Safety will be evaluated according to the NCI CTCAE Version 4.03. All observations pertinent to the safety of the study medication will be recorded on the CRF and included in the final report.
Biomarkers such as PD-L1 expression | 12 months
  The blood specimen and needle biopsy specimen would be collected

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Center Sun Yat-sen University, Guangzhou, Guangdong, China